CLINICAL TRIAL: NCT06718153
Title: Immunohistochemical Algorithm for the Diagnosis and Classification of Hepatocellular Carcinomas With TERT, TP53 and CTNNB1 Mutation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCCimmuno_2024; 2023.0275 (Other Grant/Funding Number: Fondazione Cassa di Risparmio in Bologna)
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hepatic Cancer; Hepatic Resection
Keywords: Molecular diagnostics; Immunohistochemistry
MeSH Terms: conditions — Liver Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Intervention Model Description: Diagnostic identification of possible associations between the biomarkers p53 and beta-Catenin and the presence of the genetic mutations TERT, TP53 and CTNNB1 identified by clinical practice, in patients undergoing hepatic resection of HCC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resected HCC patients (Experimental): patients resected for HCC with NGS data, and paraffin material for immunohistochemistry analysis.
  Interventions: Diagnostic Test: Immunohistochemistry and in situ hybridisation analysis

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry and in situ hybridisation analysis — immunohistochemistry and in situ hybridisation analysis for several markers, including p53, beta-Catenin and albumin, but also markers considered diagnostic for HCC such as Glutamin Synthetase, Glypican-3 and HSP70, to identify a more rational diagnostic-prognostic algorithm for primary liver lesions.

SUMMARY:
The presence of certain mutations in HCC, such as TERT and TP53, have a suspected or proven prognostic role in resected patients, but lack a morphological or immunophenotypic counterpart, which would allow us to define which tumours are rationally candidate for molecular biology analysis. The identification of a histological and immunohistochemical algorithm to determine which HCCs to take to NGS for prognostic purposes will save time and economic costs in the laboratory by rationalising available resources. In the future, the application of the immunohistochemical and molecular algorithm on biopsy could allow better prognosis and predictivity even before surgery/therapy.

DETAILED DESCRIPTION:
The primary aim is the identification of possible associations between the biomarkers p53 and beta-Catenin and the presence of the genetic mutations TERT, TP53 and CTNNB1 identified by clinical practice, in patients undergoing hepatic resection of HCC.

The secondary objective is the identification of possible associations between the presence of biomarkers Glutamin Synthetase, Glypican-3 and HSP70 and genetic mutations identified by clinical practice, in patients undergoing hepatic resection of HCC.

STUDY DESIGN: exploratory study. It is planned to recruit approximately 100 patients, who underwent liver resection for HCC and already underwent NGS analysis (for which the mutational profile is already known). All clinical and histological data will be collected, immunohistochemistry investigations will be performed on formalin-fixed and paraffin-embedded material corresponding to that used for molecular analysis.

STUDY POPULATION: The study envisages the enrolment of 100 patients, already undergoing liver resection for HCC at the IRCCS AOU of Bologna, in the period 2020-2022, who will be retrospectively re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients resected for HCC
* Availability of NGS data
* Availability of paraffin material for immunohistochemistry investigations

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
associations between p53 and beta-Catenin and the presence of the genetic mutations | At baseline
  Identification of associations between the biomarkers p53 and beta-Catenin and the presence of the genetic mutations TERT, TP53 and CTNNB1 identified by clinical practice, in patients undergoing hepatic resection of HCC.

SECONDARY OUTCOMES:
Identification of associations between the presence of biomarkers Glutamin Synthetase, Glypican-3 and HSP70 and genetic mutations | At baseline
  Identification of associations between the presence of biomarkers Glutamin Synthetase, Glypican-3 and HSP70 and genetic mutations identified by clinical practice, in patients undergoing hepatic resection of HCC.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Vasuri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No